CLINICAL TRIAL: NCT06909331
Title: Accuracy of Current Techniques in Quantifying Ketone Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRBnet: 1317538
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Placebo - Control; Exogenous Ketone Salt

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator): They were provided a placebo drink that was color, calorie and flavor-matched to the experimental drink.
  Interventions: Dietary Supplement: Placebo drink solution
- Experimental supplement (Experimental): They were provided an ketone salt drink.
  Interventions: Dietary Supplement: Exogenous ketone salt

INTERVENTIONS:
Dietary Supplement: Exogenous ketone salt — Exogenous ketone salt supplement will be taken once to determine acute circulating levels of beta-hydroxybuyrate and acetoacetate compared to a control supplement.
  Arms: Experimental supplement
Dietary Supplement: Placebo drink solution — Participants consumed a placebo drink that was flavor, color and calorie matched to the experimental drink.
  Arms: Placebo drink

SUMMARY:
The purpose of this study is to determine the accuracy of current measuring techniques used to detect physiological ketone levels.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years

Exclusion Criteria:

* taking medications that affect blood pressure, insulin, or renal function, having meta-bolic syndrome factors such as type 2 diabetes, being pregnant, and/or indicating a pre-existing health condition on the health history questionnaire

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Circulating beta-hydroxybutyrate | 30 minutes after consuming the drink
  Circulating beta-hydroxybutyrate levels measured by ketone meters and GC/MS
Circulating acetoacetate levels | 30 minutes after consuming the drink

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided